CLINICAL TRIAL: NCT02463786
Title: Improving Knowledge To Efficaciously RAise Level of Contemporary Treatment in Heart Failure
Brief Title: Improving Knowledge To Efficaciously RAise Level of Contemporary Treatment in Heart Failure (
Acronym: INTERACTinHF
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Interreg (Other)
Responsible Party: Sponsor
Other Study IDs: METC 12-4-074
Record Dates: First submitted 2015-03-16; First posted 2015-06-04 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Heart failure (HF) remains to have a poor outcome. Even though recent advances in HF led to a reduction of morbidity and mortality, improvement in outcome is much less than expected based on large randomized trials. Various reasons may be responsible, such as complexity of disease and comorbidities, inadequate diagnosis and inappropriate treatment. So far, little attention has been paid on patients seen in primary care. Also, HF care mainly focuses on the individual patient-doctor relationship. However, the increasing complexity prevents individual physicians from covering all aspects of care. Consequently, multiple stakeholders are involved, including both general practitioners and specialists. Still, the relative role, the interaction between them and the processes included are hardly defined. These aspects may not only be relevant for patient care, but also for the setup of health care systems. Whereas multidisciplinary team should resemble a seamless system across primary and hospital care, there is a scarcity of research considering how these disease management programs perform, in what form they should be offered, and what care and support patients and caregivers would benefit most.The INTERACT-in HF (Improving kNowldege Transfer to Efficaciously RAise level of Contemporary Treatment in Heart Failure) study is set up to determine and assess relevant factors of the quality of HF care. The study evaluates processes of HF care, role of relevant care givers and interactions between them. It collects data from individual patients to assess characteristics and management of contemporary HF patients. This is performed in different countries (the Netherlands, Belgium and Germany) to analyze decision making with respect to diagnostics and treatment.Cross-sectional mixed-methods are used. Patients and their caregivers are interviewed. The patient is the central starting point. Then, the treating GP, cardiologist and HF nurse are interviewed. In parallel, retrospective data based on records from these patients are reviewed to verify data from interviews and to determine characteristics of them. Retrospective data of additional patients are collected to complete the picture of the current situation. These data will be used to define bottlenecks that prevent best clinical practice to be used in daily care at all levels, comparing practice in different countries.Thus, the proposal aims to better understand HF care, which will lead to a better care and finally to improved outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients with the following inclusion criteria are suitable for participation in the study:

* age ≥18 years,
* signs, diagnosis or suspicion of heart failure and
* are contractually capable and mentally able to understand and follow the instructions of the study personnel (i.e. speaking and understanding the local language, being able to have a conversation for about an hour, being able to hear and speak).
* All subjects have to be able to give informed consent. The health care providers of these patients (cardiologists, GP's and HF-nurses) are also contacted to participate in this study.

Exclusion Criteria:

* patient who had a heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the following inclusion criteria are suitable for participation in the study: age ≥18 years, signs, diagnosis or suspicion of heart failure and are contractually capable and mentally able to understand and follow the instructions of the study personnel (i.e. speaking and understanding the local language, being able to have a conversation for about an hour, being able to hear and speak). All subjects have to be able to give informed consent. Patients who had undergone heart transplantation are excluded. Otherwise, no exclusion criteria apply. The health care providers of these patients (cardiologists, GP's and HF-nurses) are also contacted to participate in this study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of heartfailure patients characteristics in primary and secondary care | at baseline
Baseline descriptives of heart failure patients | at baseline

SECONDARY OUTCOMES:
Questionnairs: Self care behavior scale | at baseline
Questionaaire: Dutch heart failure knowlegde scale | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- MUMC, Maastricht, Netherlands